CLINICAL TRIAL: NCT05750381
Title: Assessment of Colonisation and Skin Quality Parameter Improvement by Probiotic Micrococcus Luteus Q24 Balm in Healthy Adults.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: BLIS Technologies Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: BLTCT2022/8
Record Dates: First submitted 2023-02-20; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Microbial Colonization
Keywords: probiotic
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups applying balm containing Micrococcus luteus Q24 or placebo balm.
  Group A: Probiotic Micrococcus luteus Q24 balm (dose:1e7 colony forming units per application of balm).
  Group B: Placebo balm (dose:0 colony forming units per application of balm).
Who Masked: Investigator
Masking Description: A Staff member, not part of the study group will be assigned to distribute blinded samples. The investigator will not be are of the dose groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group A: Blis Q24 balm (Active) (Active Comparator): Group A: Probiotic Micrococcus luteus Q24 balm (dose: 1e7 colony forming units per application)
  Interventions: Other: Micrococcus luteus Blis Q24 balm
- Study Group B: Placebo balm (without Blis Q24) (Placebo Comparator): Group A: Placebo balm
  Interventions: Other: Placebo balm

INTERVENTIONS:
Other: Micrococcus luteus Blis Q24 balm — Balm formulation containing probiotic bacteria Micrococcus luteus Q24 for topical applications.
  Arms: Study Group A: Blis Q24 balm (Active)
Other: Placebo balm — Placebo balm formulation for topical applications.
  Arms: Study Group B: Placebo balm (without Blis Q24)

SUMMARY:
The purpose of this study is to evaluate the skin quality improvement and colonization efficacy following the application of probiotic Micrococcus luteus Q24 (BLIS Q24) to the elbow and back of forearm in a topical balm format in healthy adults.

DETAILED DESCRIPTION:
This is a randomized double-blind, placebo-controlled pilot study with no crossover for the assessment of any changes to the microbial make-up of the skin (The local skin microbiome), detection of colonisation by the probiotic bacterium (BLIS Q24) on the skin and to evaluate the changes in skin quality parameters following topical application of probiotic in a balm format.

ELIGIBILITY:
Inclusion Criteria:

* In general good health 18 - 80 years of age.
* Practice good general body hygiene

Exclusion Criteria:

* Have a history of autoimmune disease or are immunocompromised.
* Are on concurrent antibiotic therapy or regular antibiotic use within the last 1 week.
* People with allergies or sensitivity to dairy.
* People with an open wound on the Blis Q24 application sites.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-24 (Actual); Primary Completion 2023-03-10 (Estimated); Study Completion 2023-04-12 (Estimated)

PRIMARY OUTCOMES:
Change in microbial composition on skin following application of Micrococcus luteus Q24 in balm from Day 0 (baseline) to 11 days | 11 days post intervention
  Study will determine the change in microbial composition following the application of a balm containing Micrococcus luteus Q24 balm at two body sites (elbow and back of hand). The statistical analysis will be carried out to compare the participants skin swab data from baseline to 11 days across two different sites with a level of significance of p<0.05. Overall colonization based on percentage of population colonized for different interventions will also be analyzed using appropriate statistical analysis software.
Change in microbial composition on skin following application of placebo balm from Day 0 (baseline) to 11 days | 11 days post intervention
  Study will determine the change in microbial composition following the application of a placebo balm at two body sites (elbow and back of hand). The statistical analysis will be carried out to compare the participants skin swab data from baseline to 11 days across two different sites with a level of significance of p<0.05. Overall colonization based on percentage of population colonized for different interventions will also be analyzed using appropriate statistical analysis software.
Change in microbial composition on skin post 10 days application of Micrococcus luteus Q24 in balm from Day 11 (baseline) to 18 days. | 7 days post last intervention
  Study will determine the change in microbial composition post 10 days application of Micrococcus luteus Q24 at two body sites (elbow and back of hand). The statistical analysis will be carried out to compare the participants skin swab data from Day 11 to 18 days across two different sites with a level of significance of p<0.05. Overall colonization based on percentage of population colonized for different interventions will also be analyzed using appropriate statistical analysis software.
Change in microbial composition on skin post 10 day application application of placebo balm from Day 11 (baseline) to 18 days | 7 days post last intervention
  Study will determine the change in microbial composition following the application of a placebo balm at two body sites (elbow and back of hand). The statistical analysis will be carried out to compare the participants skin swab data from Day 11 to 18 days across two different sites with a level of significance of p<0.05. Overall colonization based on percentage of population colonized for different interventions will also be analyzed using appropriate statistical analysis software.
Change in skin quality parameters following topical application Micrococcus luteus Q24 from Day 0 (baseline) to 11 days | 11 days post last intervention
  Study will determine the change in skin quality parameters using a skin quality analyzer following topical application of Micrococcus luteus Q24 balm at two body sites (elbow and back of hand). The statistical analysis will be carried out to compare the participants skin quality data from baseline to 11 days across two different sites with a level of significance of p<0.05.
Change in skin quality parameters following topical application of placebo balm from Day 0 (baseline) to 11 days | 11 days post last intervention
  Study will determine the change in skin quality parameters using a skin quality analyzer following topical application of placebo balm at two body sites (elbow and back of hand). The statistical analysis will be carried out to compare the participants skin quality data from baseline to 11 days across two different sites with a level of significance of p<0.05.
Change in skin quality parameters post 10 days application of Micrococcus luteus Q24 in balm from Day 11 (baseline) to 18 days. | 7 days post last intervention
  Study will determine the change in skin quality parameters using a skin quality analyzer following topical application of Micrococcus luteus Q24 balm at two body sites (elbow and back of hand). The statistical analysis will be carried out to compare the participants skin quality data from Day 11 to Day 18 across two different sites with a level of significance of p<0.05.
Change in skin quality parameters post 10 days application of placebo balm from Day 11 (baseline) to 18 days. | 7 days post last intervention
  Study will determine the change in skin quality parameters using a skin quality analyzer following topical application of placebo balm at two body sites (elbow and back of hand). The statistical analysis will be carried out to compare the participants skin quality data from Day 11 to Day 18 across two different sites with a level of significance of p<0.05.

CONTACTS AND LOCATIONS:
Locations (1):
- Blis Technologies Ltd, Dunedin, Otago, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Data and information in the protocol and the clinical study report will be shared to other researchers and/or in publications in due course.
Supporting Information: Study Protocol, CSR
Time Frame: Study report 3 months after completion of the study.
Access Criteria: Summary study report will be shared by the Principal Investigator upon request if not published in public literature.

REFERENCES:
- [Background] van Rensburg JJ, Lin H, Gao X, Toh E, Fortney KR, Ellinger S, Zwickl B, Janowicz DM, Katz BP, Nelson DE, Dong Q, Spinola SM. The Human Skin Microbiome Associates with the Outcome of and Is Influenced by Bacterial Infection. mBio. 2015 Sep 15;6(5):e01315-15. doi: 10.1128/mBio.01315-15. PMID 26374122
- [Background] Bourdichon F, Casaregola S, Farrokh C, Frisvad JC, Gerds ML, Hammes WP, Harnett J, Huys G, Laulund S, Ouwehand A, Powell IB, Prajapati JB, Seto Y, Ter Schure E, Van Boven A, Vankerckhoven V, Zgoda A, Tuijtelaars S, Hansen EB. Food fermentations: microorganisms with technological beneficial use. Int J Food Microbiol. 2012 Mar 15;154(3):87-97. doi: 10.1016/j.ijfoodmicro.2011.12.030. Epub 2011 Dec 31. PMID 22257932